CLINICAL TRIAL: NCT01793532
Title: Assessment of [11C]DPA-713 in Temporal Lobe Epilepsy
Brief Title: Study of [11C]DPA-713 for Temporal Lobe Epilepsy
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 130070; 13-M-0070
Record Dates: First submitted 2013-02-14; First posted 2013-02-15 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2016-07-28

CONDITIONS: Epilepsy; Temporal Lobe
Keywords: PET Imaging; Epilepsy; Inflammation; Brain Imaging
MeSH Terms: conditions — Epilepsy; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
Background:

- Some people with epilepsy have an epileptic focus, a small part of the brain that is the starting point of the seizure. This focus is like an irritant or an inflammation, and helps cause the seizure. People with epilepsy that affects the temporal lobe of the brain often have an epileptic focus. Researchers want to look at the epileptic focus by using a drug that attaches to a protein associated with inflammation. An imaging study with the drug will show how much inflammation is in the area of the brain where the seizures start. The drug, called [11C]DPA-713, will be tested for its effectiveness in people with temporal lobe epilepsy. Its effects will be compared with imaging studies given to healthy volunteers.

Objectives:

- To see if [11C]DPA-713 can show the inflammation in the epileptic focus of seizures.

Eligibility:

* Individuals at least 18 years of age who have temporal lobe epilepsy.
* Healthy volunteers at least 18 years of age.

Design:

* Participants will have three outpatient visits to the National Institutes of Health Clinical Center. The visits will last from 2 to 5 hours.
* Participants will be screened with a physical exam, neurological exam, and medical history. Blood samples will be collected before the start of the study.
* Participants will have a positron emission tomography (PET) scan. This scan will be used to look at brain chemistry and function. The study drug will be given during the scan to see how well it shows points of inflammation in the brain. Some participants will provide additional blood samples during the PET scan.
* Participants will also have a magnetic resonance imaging (MRI) scan. This scan will look at the structure of the brain.

DETAILED DESCRIPTION:
OBJECTIVE:

Translocator protein 18 kDa (TSPO) is highly expressed in activated microglia and reactive astrocytes in brain, and it may, thereby, be a useful biomarker of neuroinflammation. We developed [11C]PBR28 as a positron emission tomographic (PET) radioligand to bind to TSPO and measure its density. The purpose of this study is to assess a new TSPO radioligand, [11C]DPA-713, and to compare it with [11C]PBR28.

Although [11C]PBR28 has high in vivo specific signal, it is very sensitive to the high and low affinity states of TSPO, which are caused by a single nucleotide polymorphism (SNP) in the fourth exon of the TSPO gene. This co-dominant mutation yields three genetic groups: HH, HL, and LL, where H is the high-affinity form and L is the low affinity form. The frequency of the L allele is approximately 30%; thus, the frequency of the LL homozygote is approximately 9%. The affinity of PBR28 to H and L forms differs about 50 fold; thus, LL carriers provide no measureable signal in brain from [11C]PBR28. In contrast, the affinity of DPA-713 differs by only four-fold and LL carriers provide measureable brain uptake, although diminished in comparison to HH and HL carriers.

We recently reported that [11C]PBR28 binding is increased in epileptogenic mesial temporal lobe in HH and HL carriers, using the ratio of brain uptake in ipsilateral and contralateral regions. This study will compare [11C]DPA-713 and [11C]PBR28 in two ways. First, what is the relative robustness of absolute quantitation of TSPO in healthy subjects and patients with epilepsy, using an arterial input function and pharmacokinetic modeling? Second, what is the relative sensitivity of [11C]DPA-713 and [11C]PBR28 to detect the seizure focus in patients with epilepsy and measured as the ratio of brain uptake ipsilateral and contralateral to the seizure focus.

STUDY POPULATION

This protocol will study a total of 30 patients with epilepsy and 30 healthy human volunteers using [11C]DPA-713. Studies with [11C]PBR28 in the same subjects will be performed under other protocols, including 12-N-0182 ( Positron emission tomography measurement of neuroinflammation and P-glycoprotein in localization-related epilepsy, PI: W. Theodore).

DESIGN

For absolute quantification of TSPO, 10 patients with epilepsy and 25 healthy controls will have arterial blood sampling concurrent with PET imaging using [11C]DPA- 713. Scans of healthy subjects will also be used to study effect of the polymorphism to the binding of [11C]DPA- 713. The subjects will choose to undergo the PET scan with or without the arterial line. Most, but not all, subjects will also have a scan with [11C]PBR28 under another protocol. LL homozygotes would be excluded from [11C]PBR28 but would be included with [11C]DPA- 713.

For detection of increased TSPO receptor binding in epileptogenic foci as a ratio of ipsilateral to contralateral regions, about 20 patients with epilepsy will be studied with [11C]DPA-713. Since the ratio of brain uptake will also be obtained as part of absolute quantitation in ten patients, this ratio of brain uptake will require an additional ten subjects, who would not require an arterial catheter.

To account for dropouts and data variability, we request a ceiling of 30 epilepsy patients (about 10 of whom will have an arterial line) and 30 controls. All subjects will have blood drawn to genotype the TSPO SNP and to perform in vitro radioligand binding to TSPO on lymphocytes.

OUTCOME MEASURES

To assess absolute quantitation of TSPO with [11C]DPA-713, we will primarily use two outcome measures: the identifiability and time stability of distribution volume calculated with compartmental modeling. By comparing data of HH, HL, and LL, we will also estimate nondisplaceable distribution volume. To assess the sensitivity of [11C]DPA-713 to localize the epileptogenic focus, we will compare ratio of brain uptake in medial temporal lobe, ipsilateral and contralateral to the seizure focus.

ELIGIBILITY:
* INCLUSION CRITERIA:

For healthy volunteers

* Age 18 or older.
* Able to give written informed consent.
* No prior diagnosis of drug or alcohol abuse or dependence.

For patients

* Age 18 or older.
* Able to give written informed consent.
* Having clinically documented partial seizures with consistent EEG evidence as defined by the 1981 International Classification of Epileptic Seizures, which may be refractory or responsive to standard antiepileptic treatment. This criterion will be established by preliminary screening in the NINDS Clinical Epilepsy Section outpatient clinic under protocol 01-N-0139, and if necessary, inpatient video-EEG monitoring. Seizure focus localization will be determined by standard clinical, neurophysiologic, and imaging studies.
* Negative toxicology testing at the time of screening.
* No prior diagnosis of drug or alcohol abuse or dependence.

EXCLUSION CRITERIA:

For healthy volunteers

* Any current Axis I diagnosis.
* Clinically significant laboratory abnormalities.
* Positive test for HIV.
* Unable to have a MRI scan.
* History of neurologic illness or injury with the potential to affect study data interpretation.
* History of seizures, other than in childhood and related to fever.
* Recent exposure to radiation (i.e., PET from other research) which when combined with this study would be above the allowable limits.
* Inability to lie flat on camera bed for at least two hours.
* Pregnancy or breast feeding.
* Able to get pregnant but does not use birth control.
* Drug/alcohol abuse or dependence

For patients

* Previous radiation exposure (X-rays, PET scans etc.) that, together with study procedures, would exceed NIH RSC research limits.
* Claustrophobia to a degree that the subject would feel uncomfortable in the MRI machine.
* History of brain disease other than epilepsy.
* Cannot lie on their back for at least two hours.
* Known cause for seizures, other than mesial temporal sclerosis, such as tumor or infection.
* Serious medical illness, other than epilepsy.
* Clinically significant laboratory abnormalities.
* Positive test for HIV.
* Brain abnormality such as a brain tumor, stroke, brain damage from head trauma or blood vessel abnormalities, on an MRI scan.
* Pregnancy or breast feeding.
* Able to get pregnant but does not use birth control.
* Risk for MRI scan, such as a pacemaker or other implanted electrical devices, brain stimulators, some types of dental implants, aneurysm clips (metal clips on the wall of a large artery), metallic prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, implanted delivery pump, or shrapnel fragments. Welders and metal workers are also at risk for injury because of possible small metal fragments in the eye of which they may be unaware.
* For drug-responsive subjects: occurrence of a seizure within the last three months.
* Drug/alcohol abuse or dependence

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-01-31; Primary Completion 2016-06-08 (Actual); Study Completion 2016-06-08 (Actual)

PRIMARY OUTCOMES:
Brain uptake of radioligand | 90 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Innis, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Boutin H, Chauveau F, Thominiaux C, Gregoire MC, James ML, Trebossen R, Hantraye P, Dolle F, Tavitian B, Kassiou M. 11C-DPA-713: a novel peripheral benzodiazepine receptor PET ligand for in vivo imaging of neuroinflammation. J Nucl Med. 2007 Apr;48(4):573-81. doi: 10.2967/jnumed.106.036764. PMID 17401094
- [Background] Banati RB, Newcombe J, Gunn RN, Cagnin A, Turkheimer F, Heppner F, Price G, Wegner F, Giovannoni G, Miller DH, Perkin GD, Smith T, Hewson AK, Bydder G, Kreutzberg GW, Jones T, Cuzner ML, Myers R. The peripheral benzodiazepine binding site in the brain in multiple sclerosis: quantitative in vivo imaging of microglia as a measure of disease activity. Brain. 2000 Nov;123 ( Pt 11):2321-37. doi: 10.1093/brain/123.11.2321. PMID 11050032
- [Background] Banati RB, Myers R, Kreutzberg GW. PK ('peripheral benzodiazepine')--binding sites in the CNS indicate early and discrete brain lesions: microautoradiographic detection of [3H]PK11195 binding to activated microglia. J Neurocytol. 1997 Feb;26(2):77-82. doi: 10.1023/a:1018567510105. PMID 9181482